CLINICAL TRIAL: NCT02218983
Title: The Prognostic Value of Limited Transthoracic Echocardiogram (LTTE) During Trauma Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Principal Investigator, Aron Depew, MD, Principal Investigator, Riverside University Health System Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 620651
Record Dates: First submitted 2014-08-01; First posted 2014-08-18 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Patients Who Are in Shock and Intubated in the Trauma Bay (TB)
Keywords: trauma; echo; echocardiogram; ultrasound; inferior vena cava collapsibility
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Limited transthoracic echocardiogram (LTTE) (Experimental): LTTE (SonoSite Ultrasound), which will be performed every 10 - 30 minutes, after each fluid challenge or transfusion, until two consecutive equivalent measurements are reached without fluid challenge or transfusion
  Interventions: Device: Limited Transthoracic Echocardiogram (LTTE, SonoSite Ultrasound)
- Usual care (Active Comparator): measurements on :blood pressure, heart rate, urine output, lactate, lactate clearance (after 6 hrs), base deficit, creatinine
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Limited Transthoracic Echocardiogram (LTTE, SonoSite Ultrasound)
  Arms: Limited transthoracic echocardiogram (LTTE)
Other: Usual care
  Arms: Usual care

SUMMARY:
Primary caregiver thoracic ultrasound (U/S) is a skill which is growing in utility in critical care. First introduced for volume assessment in nephrology and cardiology, it is now being researched in emergency and critical care. Data is still evolving in its use in initial trauma evaluation. Inferior vena cava (IVC) diameter correlates with outcome in trauma, but utility of its measurement on U/S in the emergency department still has some controversy. In trauma specifically, small studies suggests benefit to the use of U/S to predict volume status, and most of these data are from one author. It is not known if this can be applied more broadly. The prognostic value of findings on limited transthoracic echocardiogram (LTTE, SonoSite Ultrasound) has been studied in several small studies, and only one small randomized controlled trial has proven benefit to its use. Due to inter-rater reliability and the fact that all reports on credentialing of thoracic ultrasound use in the trauma bay are from one group, it is not known if it can be applied to all trauma populations.

Research question:

Does LTTE (SonoSite Ultrasound) predict mortality, emergency surgery, intensive care unit (ICU) stay, hospital stay, time on ventilator, number of transfusions, or renal failure as well as or better than other methods of organ perfusion?

Hypotheses:

1. Use of LTTE is associated with improved outcomes (less organ failure, decreased hospital and ICU stays, transfusions, and mortality).
2. LTTE predicts mortality, emergency surgery, ICU stay, hospital stay, time on ventilator, number of and transfusions better than other methods of organ perfusion (tachycardia, hypotension, lactate, lactate clearance, creatinine, base deficit).

ELIGIBILITY:
Inclusion Criteria:

* Patients arriving to trauma bay aged 18 or higher
* Hypotensive (systolic blood pressure (SBP) < 90 mmHg or mean arterial pressure (MAP) < 65, on 2 measurements)
* Respiratory failure (requiring mechanical ventilation)

Exclusion Criteria:

* Unable to draw blood before transfusion or fluid challenge
* Patient arrests within 10 minutes of arrival
* Pregnant

Note: If inferior vena cava (IVC) not visible on ultrasound (U/S), pt will go to non-IVC group.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
length of stay in the intensive care unit | length of stay in the intensive care unit, not to exceed 30 days

SECONDARY OUTCOMES:
mortality (death) | mortality (death) during hospital stay, not to exceed 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Aron Depew, MD, Principal Investigator — Riverside University Health System Medical Center
Locations (1):
- Riverside County Regional Medical Center, Moreno Valley, California, United States